CLINICAL TRIAL: NCT04776369
Title: Effect of Intravenous Single-bolus Lidocaine Infusion Versus Intravenous Single-bolus Magnesium Sulfate Infusion on Postoperative Pain, Emotional Status and Quality of Life in Patients Undergoing Spine Fusion Surgery
Brief Title: Effect of Lidocaine Versus Magnesium on Postoperative Pain in Spine Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Haitham Mohammad Ahmad Mohammad (Other)
Responsible Party: Sponsor-Investigator, Haitham Mohammad Ahmad Mohammad, Principal investigator, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Pain after spine fusion
Record Dates: First submitted 2021-02-23; First posted 2021-03-01 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Magnesium Sulfate; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to 4 groups:
  * Group A: 30 patients will receive IV lidocaine 4 mg/kg (Tan, 2019) in 50 ml volume over 30 min. plus IV saline 50 ml after induction of anesthesia.
  * Group B: 30 patients will receive IV magnesium sulfate 30mg/kg in 50 ml volume over 30 min. plus IV saline 50 ml after induction of anesthesia.
  * Group C: 30 patients will receive IV lidocaine 4 mg/kg in 50 ml volume over 30 min. plus IV magnesium sulfate 30mg/kg in 50 ml volume over 30 min. after induction of anesthesia.
  * Group D (control group): 30 patients will receive IV saline 50 ml plus IV saline 50 ml over 30 min. after induction of anesthesia.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Lidocaine group (Active Comparator): 30 patients will receive IV lidocaine 4 mg/kg in 50 ml volume over 30 min. plus IV saline 50 ml after induction of anesthesia.
  Interventions: Drug: Lidocaine IV; Drug: IV saline
- Magnesium group (Active Comparator): 30 patients will receive IV magnesium sulfate 30 mg/kg in 50 ml volume over 30 min. plus IV saline 50 ml after induction of anesthesia.
  Interventions: Drug: Magnesium Sulfate Injection; Drug: IV saline
- Combination group (Active Comparator): 30 patients will receive IV lidocaine 4 mg/kg in 50 ml volume over 30 min. plus IV magnesium sulfate 30 mg/kg in 50 ml volume over 30 min. after induction of anesthesia.
  Interventions: Drug: Lidocaine IV; Drug: Magnesium Sulfate Injection
- control group (Placebo Comparator): 30 patients will receive IV saline 50 ml plus IV saline 50 ml over 30 min. after induction of anesthesia.
  Interventions: Drug: IV saline

INTERVENTIONS:
Drug: Lidocaine IV — single-bolus of lidocaine IV 4 mg/kg
  Arms: Combination group; Lidocaine group
Drug: Magnesium Sulfate Injection — single-bolus of magnesium sulfate IV 30 mg / kg
  Arms: Combination group; Magnesium group
Drug: IV saline — Saline IV 50 ml
  Arms: Lidocaine group; Magnesium group; control group

SUMMARY:
The goal in this work is to compare the effect of intravenous single-bolus lidocaine infusion versus intravenous single-bolus magnesium sulfate infusion on postoperative pain, emotional status and quality of life in patients undergoing spine fusion surgery.

DETAILED DESCRIPTION:
This is a double-blinded prospective controlled randomized clinical trial that will be performed in Assiut university hospital.

After obtaining approval from Assiut University Hospital Ethical Committee and informed written consent from patients, this study will be conducted on ASA status I, II and III patients, aged between 18y and 60 y, both male and female, undergoing spinal fusion surgery (single, and double level).

Subjects will be excluded if they met any of the following criteria: Previous spine surgery, morbid obesity (BMI > 40), spine metastatic tumor, allergy to an amide LA, or magnesium sulfate, heart block, renal, or liver dysfunction, substance abuse disorder, chronic opioid use, or electrolyte disturbance , administration of any sedative, preexisting mental illness, psychological or emotional problems.

Randomization will be performed using lidocaine group, magnesium group, combined (lidocaine and magnesium) group and control group registers, which will be placed in sealed envelopes prior to study initiation, and opened prior to anesthesia by a physician who will prepare the IV solution, and identify it with the patient number, according to the envelope drawn. The solution will be handed to another physician, blind to the prepared solutions' content, who will be responsible for the anesthesia. The solution volume will be equal. The responsible investigator will remain blind to the chosen group until the end of the study.

Allocation concealment will be done using serially numbered closed, opaque envelopes. Each patient will be given a serial number from a computer-generated randomization table, and will be placed in the appropriate group after opening the corresponding sealed envelope. Counseling for participation will be conducted before recruitment.

Operative technique: Patients will be monitored with continuous electrocardiography, capnography, pulse oximetry, and intermittent non-invasive blood pressure measurements every 5 minutes.

After establishment of venous access, anesthesia will be induced with propofol 2 mg / kg, fentanyl 1.5 µg / kg and cisatracurium 0.15 mg/kg. Endotracheal tube of appropriate size will be inserted and mechanical ventilation utilizing isoflurane in oxygen/air mixture at sufficient concentration to maintain systolic blood pressure within the limit of 20% baseline value.

All patients will receive 30 mg ketorolac IV infusion after induction of anesthesia, Paracetamol 1g will be given by IV infusion to all patients before extubation. Reversal of residual muscle relaxant will be accomplished using neostigmine, and atropine at the end of the operation guided by train of four.

Intraoperative fluid therapy will be administered in the form of normal saline after calculation of fasting and maintenance fluid requirements.

Patients will be discharged to PACU then to the ward after fulfilling the standard criteria.

No other anesthetics or sedatives will be allowed during the operation. In the first 24 hours postoperative; patients will be given Ketorolac 30 mg slowly IV (diluted to 10 ml) every 12h, and paracetamol 1g injection every 8 hours; starting 8 hours after extubation. Morphine 0.1mg/kg slowly IV will be given as rescue analgesia when numeric rating scale (NRS) is ≥4, or if the patient requested additional analgesia, with a minimum 8 hours interval between the 2 consecutive injections. Total doses of IV morphine will be documented.

After 24 hours post-operation; paracetamol 1 g every 8 hours will be given orally for 5 days. Ketolac 30 mg will be given orally only if needed.

Pain will be assessed during rest and cough in the first 24 h, and during movement after 24h. postoperative.

All patients will be urged to ambulate as early as practically possible. Collected data will include patient's characteristics, and surgical data including age, gender, weight, height, duration of surgery, and duration of hospital stay. Postoperative pain evaluation during rest will be assessed by numeric rating scale (NRS). Patients' satisfaction will be assessed by using 5 points Likert score for satisfaction where 1=strongly dissatisfied; 2=Dissatisfied; 3=neither satisfied nor dissatisfied; 4=Satisfied; 5=strongly satisfied. The two scores will be recorded at the following times: immediately at 1 h; 6 h; 12 h; 24 h; at discharge time; 1 month; 2 months, and 3 months postoperative.

Time to the first request for analgesia and the total dose of rescue analgesia (morphine) in the first 24 hours after surgery will be recorded. The long-term follow-up of postoperative back pain for 3 months will be conducted through the outpatient orthopedic clinic, or by telephone.

Hemodynamics and blood loss will be reported First time to pass flatus, first time to defecate and incidence of complications will also be reported (such as hypotension, bradycardia, anxiety, dizziness, muscle twitching, nervousness, reaction at the site of injection, cardiac arrest, double vision, nausea, seizures, unconsciousness, euphoria, tinnitus, vomiting).

Testing for gross mental and neurologic defects will be performed with the Mini-Mental Status Examination, which has a standard scoring method with a maximum score of 30. The total duration of the testing will not exceed 45 minutes. Interruptions will be allowed at the request of the patient between, but not within, individual tests of the session. The tests will be administered by the same examiner to limit interexaminer variability.

The anxiety and depression status will be evaluated by Self-Rating Anxiety Scale (SAS) and Self-Rating Depression Scale (SDS), and QOL will be measured by Short Form Health Survey 36 (SF-36) in eight sections, including vitality, physical functioning, bodily pain, general health perceptions, mental health, physical, emotional, and social role functioning.

The study portion of the tests will be performed at least 6 hours after the initial intravenous bolus of drugs, while the control portion will be performed at least 24 hours after the studied drugs are discontinued. Tests will be repeated after 1 week and 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* ASA status I, II and III patients
* Age 18 - 60 y
* Gender: both male and female
* Undergoing spinal fusion surgery (single, and double level).

Exclusion Criteria:

* Previous spine surgery
* Morbid obesity (BMI > 40)
* Spine metastatic tumor
* Allergy to an amide LA, or magnesium sulfate
* Heart block, renal, or liver dysfunction
* Substance abuse disorder, or chronic opioid use, administration of any sedative or preexisting mental illness.
* Electrolyte disturbance.
* Psychological or emotional problems.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
short-term postoperative pain control | first 24 hours postoperative (Day 0)
  Short-term pain control will be assessed in the first 24 hours postoperative. by numeric rating scale (NRS). It ranges from 0 to 10 where 0= no pain and 10= maximum pain

SECONDARY OUTCOMES:
long-term pain control | Every month till 3 months (Month 1, Month 2, Month 3)
  long-term pain control will be assessed by numeric rating scale (NRS), It ranges from 0 to 10 where 0= no pain and 10= maximum pain
Total opioid consumption | Every month till 3 months (Month 1, Month 2, Month 3)
  Total opioid consumption will be calculated
Mental state, Anxiety and depression , quality of life | 6 hours postoperative, 24 hours postoperative, 1 week postoperative, 4 weeks postoperative
  Mini-mental state scale, Self-rating anxiety scale (SAS), Self-rating depression scale (SDS) and short form health survey 36 scale(SF-36).

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Albrecht E, Kirkham KR, Liu SS, Brull R. Peri-operative intravenous administration of magnesium sulphate and postoperative pain: a meta-analysis. Anaesthesia. 2013 Jan;68(1):79-90. doi: 10.1111/j.1365-2044.2012.07335.x. Epub 2012 Nov 1. PMID 23121612
- [Result] Amir R, Argoff CE, Bennett GJ, Cummins TR, Durieux ME, Gerner P, Gold MS, Porreca F, Strichartz GR. The role of sodium channels in chronic inflammatory and neuropathic pain. J Pain. 2006 May;7(5 Suppl 3):S1-29. doi: 10.1016/j.jpain.2006.01.444. PMID 16632328
- [Result] Apfelbaum JL, Chen C, Mehta SS, Gan TJ. Postoperative pain experience: results from a national survey suggest postoperative pain continues to be undermanaged. Anesth Analg. 2003 Aug;97(2):534-540. doi: 10.1213/01.ANE.0000068822.10113.9E. PMID 12873949
- [Result] Dunn LK, Yerra S, Fang S, Hanak MF, Leibowitz MK, Tsang S, Durieux ME, Nemergut EC, Naik BI. Incidence and Risk Factors for Chronic Postoperative Opioid Use After Major Spine Surgery: A Cross-Sectional Study With Longitudinal Outcome. Anesth Analg. 2018 Jul;127(1):247-254. doi: 10.1213/ANE.0000000000003338. PMID 29570151
- [Result] Gupta K, Vohra V, Sood J. The role of magnesium as an adjuvant during general anaesthesia. Anaesthesia. 2006 Nov;61(11):1058-63. doi: 10.1111/j.1365-2044.2006.04801.x. PMID 17042843
- [Result] Kosharskyy B, Almonte W, Shaparin N, Pappagallo M, Smith H. Intravenous infusions in chronic pain management. Pain Physician. 2013 May-Jun;16(3):231-49. PMID 23703410
- [Result] Kim KT, Cho DC, Sung JK, Kim YB, Kang H, Song KS, Choi GJ. Intraoperative systemic infusion of lidocaine reduces postoperative pain after lumbar surgery: a double-blinded, randomized, placebo-controlled clinical trial. Spine J. 2014 Aug 1;14(8):1559-66. doi: 10.1016/j.spinee.2013.09.031. Epub 2013 Nov 8. PMID 24216403
- [Result] Lenart MJ, Wong K, Gupta RK, Mercaldo ND, Schildcrout JS, Michaels D, Malchow RJ. The impact of peripheral nerve techniques on hospital stay following major orthopedic surgery. Pain Med. 2012 Jun;13(6):828-34. doi: 10.1111/j.1526-4637.2012.01363.x. Epub 2012 Apr 11. PMID 22494645